CLINICAL TRIAL: NCT03502135
Title: Efficacy of Tetracaine/Oxymetazoline Nasal Spray for Endodontic Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study drug not available in time
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0417
Record Dates: First submitted 2018-03-22; First posted 2018-04-18 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Endodontic Disease; Endodontic Inflammation; Local Anesthesia; Dental Anesthesia
MeSH Terms: conditions — Dental Pulp Diseases; Pulpitis | interventions — Tetracaine

STUDY DESIGN:
Intervention Model Description: Single-Arm, unblinded trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intranasal Anesthesia (Experimental): Two intranasal sprays of tetracaine HCl and oxymetazoline HCl nasal spray anesthetic administered 4 minutes apart into the nostril corresponding to the side of the treated tooth. If inadequate anesthetic response obtained within 10 minutes, a third spray will be administered and assessed for effective anesthesia after 4 minutes.
  Interventions: Drug: Tetracaine HCl and oxymetazoline HCl nasal spray

INTERVENTIONS:
Drug: Tetracaine HCl and oxymetazoline HCl nasal spray — Two intranasal sprays of anesthetic. Each spray delivers 0.2 mL of solution containing 6 mg tetracaine hydrochloride and 0.1 mg of oxymetazoline hydrochloride

SUMMARY:
Purpose:

To evaluate anesthetic efficacy and overall patient experience with use of Kovanaze tetracaine/oxymetazoline nasal spray for root canal treatment of vital premolar and anterior teeth needing root canal treatment.

Participants:

30 adult patients with a vital upper anterior or premolar tooth (#4-13) with a diagnosis indicating need root canal treatment and who are seeking treatment in the UNC Chapel Hill School of Dentistry.

Procedures (methods):

Qualifying patients will be anesthetized with tetracaine/oxymetazoline nasal spray anesthetic in order to facilitate completion of their clinically required, standard of care root canal treatment. Research procedures include blood pressure monitoring and pain assessment using a visual analogue pain scale.

DETAILED DESCRIPTION:
The study will be undertaken in the UNC Chapel Hill School of Dentistry student clinics. Eligible patients seeking treatment at the School of Dentistry will be recruited to the study and written informed consent obtained.

Operator Training:

Operators will obtain online and in person training to ensure consistent, accurate use of the nasal spray. Anesthesia of all study subjects will be performed by UNC Chapel Hill Graduate Endodontics residents.

Patient Selection:

A total of thirty adult subjects (>18years old) seeking endodontic treatment will be recruited to the study. Inclusion criteria are: American Society of Anesthesiologists class I or II; Preoperative heart rate of 55 to 100 beats per minute; a maximum blood pressure reading of 166/100 mmHg; maxillary anterior tooth or premolar with a diagnosis or treatment plan which indicates root canal treatment.

Exclusion criteria are based on recommendations made by the FDA label as well the adverse effects reported in prior clinical trials.

History, examination, and recruitment:

Information including history of present illness, vital signs (heart rate and blood pressure) and medical history will be obtained. Standardized, calibrated examiners will perform a standard endodontic clinical exam including the response to cold ascertained using a cold stimulus (EndoIce, Coltène/Whaledent, Cuyahoga Falls, OH). Written informed consent will be obtained from patients who meet the study criteria and agree to participate.

Participating patients will be asked to rate their current pain on a 100 mm Visual Analogue Scale. No pain will correspond to 0 mm, mild pain as less than 30 mm, moderate to severe pain from 30 to 100 mm.

Anesthesia:

Two intranasal sprays of anesthetic (each spray 6mg tetracaine HCl, 0.1mg oxymetazoline) will be administered 4 minutes apart on the side of the tooth to be treated. After an interval of 10 minutes, pulpal anesthesia will be ascertained by re-evaluating pain level with the VAS scale, as well as application of a cold stimulus. If adequate pulpal anesthesia is noted, the operator will commence with treatment. If the patient has a positive response to cold stimulus on the tooth or a persisting spontaneous moderate to severe pain on the VAS, then a third spray of tetracaine/oxymetazoline will be administered. After a time interval of 4 minutes the operator will again test for pulpal anesthesia. If at this point pulpal anesthesia is not noted then the failure to obtain adequate anesthesia will be recorded and rescue anesthesia will be provided. Root canal treatment will be initiated immediately once pulpal anesthesia has been ascertained. A timer will be started at this point in order to record any subsequent time of failure.

Treatment:

The tooth will be isolated with a rubber dam and the pulp chamber will be accessed with a high-speed dental handpiece. Standard root canal treatment will subsequently be initiated and performed. If at any point during treatment the patient feels pain, the procedure will be stopped and pain intensity will be assessed via the aforementioned VAS pain scale. A reported moderate to severe pain score will necessitate additional anesthetic. The stage and time after initiation of treatment that pain occurred (access, instrumentation, or obturation) will be recorded. After three tetracaine/oxymetazoline sprays, rescue anesthesia will be administered if a moderate to severe pain score persists.

Success will be defined as ability to perform complete cleaning and shaping of the tooth's root(s). If additional rescue anesthesia is required at any point in during treatment, the nasal spray anesthesia will be considered a failure. If rescue anesthesia is required during subsequent stages of treatment, the stage will be recorded for subjective documentation.

Data Analysis:

An exact binomial test with a nominal 0.05 two-sided significance level will have 93% power to detect the difference between the null hypothesis proportion of 0.5 (random chance) and the alternative proportion of 0.8 when the sample size is 30. Secondary analysis will evaluate the proportion of patients that demonstrated sufficient pulpal anesthesia to commence treatment. For patients who required rescue anesthesia, the stage of treatment and time until rescue was needed will be analyzed. The success rate of premolars vs. anterior teeth will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I or II
* Preoperative heart rate of 55 to 100 beats per minute
* Maximum blood pressure reading of 166/100 mmHg
* Maxillary anterior tooth or premolar with a diagnosis or treatment plan which indicates root canal treatment

Exclusion Criteria:

* Inadequately controlled thyroid disease
* Five or more nosebleeds in the past month
* Known allergy to any study drug or para-aminobenzoic acid
* History of methemoglobinemia
* Taking monoamine oxidase inhibitors, tricyclic antidepressants (i.e. amitriptyline), or non-selective beta adrenergic antagonists (i.e. propranolol);
* Taking oxymetazoline-containing products (i.e., Afrin) in the last 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that are successfully anesthetized for endodontic treatment | From beginning to end of endodontic treatment appointment (about 1 to 1.5 hours)
  Anesthetic success is defined as having sufficiently anesthetize teeth to allow for endodontic treatment.

SECONDARY OUTCOMES:
Proportion of patients demonstrating sufficient pulpal anesthesia to commence treatment | From beginning to end of endodontic treatment appointment (about 1 to 1.5 hours)
Stage of anesthesia failure | From beginning to end of endodontic treatment appointment (about 1 to 1.5 hours)
  Evaluation of treatment stage (if any) at which anesthesia fails. Progressive stages at which failure may occur include 1. After Anesthesia 2. While cutting into dentin 3. Upon access of the pulp 4. Upon instrumentation of the canals
Proportion of premolars vs. anterior teeth successfully anesthetized | From beginning to end of endodontic treatment appointment (about 1 to 1.5 hours)
  Anesthesia success rate of vital premolars vs. anterior teeth receiving treatment will be compared
Time of anesthesia failure after completion of anesthetic administration | From administration of anesthesia to completion of endodontic treatment appointment (about 1 hour)

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khan, DDS, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No